CLINICAL TRIAL: NCT04493619
Title: A Multicenter, Open-Label, Parallel, Phase 2a Study of PLX2853 Monotherapy in Advanced Gynecological Malignancies With a Known ARID1A Mutation and Phase 1b/2a Study of PLX2853/Carboplatin Combination Therapy in Platinum-Resistant Epithelial Ovarian Cancer
Brief Title: PLX2853 as a Single Agent in Advanced Gynecological Malignancies and in Combination With Carboplatin in Platinum-Resistant Epithelial Ovarian Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: study terminated due to business realignment
Sponsor: Opna Bio LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PLX124-03
Record Dates: First submitted 2020-07-23; First posted 2020-07-30 (Actual); Results first posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Gynecologic Neoplasms; Epithelial Ovarian Cancer
Keywords: PLX2853; Ovarian Cancer; ARID1A; Gynecological Malignancies; Carboplatin
MeSH Terms: conditions — Genital Neoplasms, Female; Carcinoma, Ovarian Epithelial; Ovarian Neoplasms | interventions — Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 2a PLX2853 Monotherapy (80 mg) (Experimental): Subjects with ARID1A mutation-positive advanced gynecological malignancies
  Interventions: Drug: PLX2853
- Phase 1b PLX2853 (40 mg) + Carboplatin Combination Therapy (Experimental): Subjects with platinum-resistant EOC
  Interventions: Drug: PLX2853; Drug: Carboplatin
- Phase 2a PLX2853 (80 mg) + Carboplatin Combination Therapy (Experimental): Subjects with platinum-resistant EOC
  Interventions: Drug: PLX2853; Drug: Carboplatin
- Phase 1b PLX2853 (80 mg) + Carboplatin Combination Therapy (Experimental): Subjects with platinum-resistant EOC
  Interventions: Drug: PLX2853; Drug: Carboplatin

INTERVENTIONS:
Drug: PLX2853 — PLX2853 tablets
Drug: Carboplatin — Carboplatin IV injection, 5 mg•min/mL
  Arms: Phase 1b PLX2853 (40 mg) + Carboplatin Combination Therapy; Phase 1b PLX2853 (80 mg) + Carboplatin Combination Therapy; Phase 2a PLX2853 (80 mg) + Carboplatin Combination Therapy

SUMMARY:
The purpose of this research study is to evaluate safety, pharmacokinetics, pharmacodynamics and preliminary efficacy of the investigational drug PLX2853 in Advanced Gynecological Malignancies with a Known ARID1A Mutation and PLX2853/Carboplatin Combination Therapy in Platinum-Resistant Epithelial Ovarian Cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the time of signing informed consent
2. Histologically or cytologically confirmed diagnosis of 1 of the following, and must have measurable disease per RECIST v1.1:

   * Phase 2a (PLX2853 monotherapy): Any advanced gynecological malignancy (cervical, vaginal, vulvar, uterine, ovarian, fallopian tube, or primary peritoneal) with a known ARID1A mutation, that is intolerant to or refractory to all standard therapy known to confer clinical benefit.
   * Phase 1b and Phase 2a (PLX2853 + carboplatin combination):

   Platinum-resistant EOC (including fallopian tube or primary peritoneal cancer).
3. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to 1
4. Adequate organ function as demonstrated by laboratory values.
5. Women of child bearing potential (defined as any female who has experienced menarche and who has not undergone successful surgical sterilization or is not postmenopausal) must have a negative serum pregnancy test within 7 days prior to taking the first dose of study drug and, if sexually active, must agree to use a highly effective method of contraception (a contraception method with a failure rate <1% per year) and 1 additional barrier method from the time of the negative pregnancy test to 90 days after the last dose of study drug. Women of non-child bearing potential may be included if they are either surgically sterile or have been postmenopausal for ≥1 year.
6. Except as specified above for organ function, all drug-related toxicity from previous cancer therapy must be resolved (to Grade ≤1 or baseline per National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 [NCI CTCAE v5.0]) prior to study treatment administration (Grade 2: alopecia, hot flashes, decreased libido, or neuropathy is allowed).
7. Willingness and ability to provide written informed consent prior to any study-related procedures and to comply with all study requirements

Exclusion Criteria:

1. Prior exposure to a bromodomain inhibitor
2. Ongoing systemic infection requiring treatment with antibiotic, antiviral, or antifungal treatment
3. Autoimmune hemolytic anemia or autoimmune thrombocytopenia
4. Presence of symptomatic or uncontrolled central nervous system or leptomeningeal metastases
5. Red blood cell or platelet transfusion within 14 days of Screening blood draw
6. Known or suspected allergy to the investigational agent or any agent given in association with this study
7. Use of biotin (i.e., Vitamin B7) or supplements containing biotin higher than the daily adequate intake of 30 μg (NIH-ODS 2020).
8. Use of strong inhibitors and inducers of CYP3A4 and 2C8
9. Clinically significant cardiac disease
10. Inability to take oral medication or significant nausea and vomiting, malabsorption, or significant small bowel resection that, in the opinion of the Investigator, would preclude adequate absorption
11. Non-healing wound, ulcer, or bone fracture
12. Infection with HIV-1 or HIV-2. Exception: subjects with well-controlled HIV (e.g., CD4 >350/mm3 and undetectable viral load) are eligible.
13. Current active liver disease from any cause, including hepatitis A (hepatitis A virus immunoglobulin M positive), hepatitis B (hepatitis B virus [HBV] surface antigen positive), or hepatitis C (hepatitis C virus [HCV] antibody positive, confirmed by HCV ribonucleic acid).
14. Active known second malignancy with the exception of any of the following:

    * Adequately treated basal cell carcinoma, squamous cell carcinoma of the skin, or in situ cervical cancer
    * Adequately treated Stage I cancer from which the subject is currently in remission and has been in remission for ≥2 years
    * Any other cancer from which the subject has been disease-free for ≥3 years
15. Major surgery or significant traumatic injury within 28 days prior to Cycle 1 Day 1
16. Hospitalization for subacute bowel obstruction within 28 days prior to Cycle 1 Day 1
17. Receipt of anti-cancer therapy prior to Cycle 1 Day 1:

    * Chemotherapy, radiation therapy, or small molecule anti-cancer therapy for the treatment of cancer within 14 days or 5 half-lives (whichever is shorter) of Cycle 1 Day 1
    * Immune therapy or other biologic therapy (e.g., monoclonal antibodies, antibody-drug conjugates) for the treatment of cancer within 21 days or 5 half-lives (whichever is shorter) of Cycle 1 Day 1 Subjects can receive a stable dose of bisphosphonates for bone metastases, before and during the study as long as these were started at least 28 days prior to treatment with study drug.
18. Subject is participating in any other therapeutic clinical study (observational or registry studies are allowed).
19. Subjects who are pregnant or breast-feeding
20. Presence of any other medical, psychological, familial, sociological, or geographic condition potentially hampering compliance with the study protocol or would interfere with the study endpoints or the subject's ability to participate.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (8):
  - The University of Chicago Medical Center, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Oklahoma - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Tennessee Oncology / Sarah Cannon, Nashville, Tennessee
  - University of Virginia Health Systems, Charlottesville, Virginia
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - University of Washington / Seattle Cancer Care Alliance, Seattle, Washington
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 2a: PLX2853 80 mg once/day monotherapy
- Phase 1b Combination; Phase 2a Combination: PLX2853 40 mg once/daily + carboplatin once every 28 days
- Phase 1b: PLX2853 80 mg once/daily + carboplatin once every 28 days
Period: Overall Study
Arm/Group | Phase 2a | Phase 1b Combination | Phase 1b | Phase 2a Combination
Started | 14 | 3 | 7 | 13
Completed | 0 | 0 | 0 | 0
Not Completed | 14 | 3 | 7 | 13
Not completed — Death | 4 | 3 | 3 | 4
Not completed — Study discontinued early | 10 | 0 | 4 | 8
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- PLX2853 Phase 2a Monotherapy: Up to 26 evaluable subjects with ARID1A mutation-positive advanced gynecological malignancies will be enrolled.
  PLX2853: PLX2853 tablets
- PLX2853 (40 mg) + Carboplatin Phase 1b; PLX2853 (80 mg) + Carboplatin Phase 1b: Phase 1b (PLX2853 + carboplatin combination): Up to 15 evaluable subjects with platinum-resistant EOC will be enrolled.
  PLX2853: PLX2853 tablets
  Carboplatin: Carboplatin IV injection, 5 mg•min/mL
- PLX2853 + Carboplatin Phase 2a Combination Therapy: Phase 2a (PLX2853 + carboplatin combination): Up to 26 evaluable subjects with platinum-resistant EOC will be enrolled.
  PLX2853: PLX2853 tablets
  Carboplatin: Carboplatin IV injection, 5 mg•min/mL
- Total: Total of all reporting groups
Arm/Group | PLX2853 Phase 2a Monotherapy | PLX2853 (40 mg) + Carboplatin Phase 1b | PLX2853 (80 mg) + Carboplatin Phase 1b | PLX2853 + Carboplatin Phase 2a Combination Therapy | Total
Number analyzed (Participants) | 14 | 3 | 7 | 13 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 2 | 4 | 9 | 25
  >=65 years | 4 | 1 | 3 | 4 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 3 | 7 | 13 | 37
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 0 | 11 | 14
  Not Hispanic or Latino | 9 | 3 | 5 | 0 | 17
  Unknown or Not Reported | 2 | 0 | 2 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 2 | 0 | 4
  White | 11 | 1 | 4 | 11 | 27
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 0 | 0 | 3
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 0 | 0 | 3 | 3
  United States | 14 | 0 | 7 | 10 | 34

OUTCOME MEASURES:

1. Primary Outcome: Phase 2a (PLX2853 Monotherapy): Number of Participants With Overall Response Rate (ORR) as Measured by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: Overall response rate as measured by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Time Frame: From 8 weeks of treatment for only PLX2853 (Cycle 3 Day 1; 28 days per cycle) until completion of long term follow-up, an average of 6 months.
Population: This outcome measure was not evaluated. The study was discontinued early and continued collection of disease status, which is required to determine overall response rate (ORR), was not conducted, therefore this measure is not reportable.
Groups:
- PLX2853 Phase 2a Monotherapy: Subjects with ARID1A mutation-positive advanced gynecological malignancies will be enrolled.
- PLX2853 + Carboplatin Phase 1b/2a Combination Therapy: Subjects with platinum-resistant EOC
Arm/Group | PLX2853 Phase 2a Monotherapy | PLX2853 + Carboplatin Phase 1b/2a Combination Therapy
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Phase 1b (PLX2853 + Carboplatin Combination): Establish the Number of Participants Reaching MTD/RP2D for the Combination of PLX2853 and Carboplatin
Description: MTD is defined as the maximum tolerated dose, which is determined from dose-limiting toxicity. If DLTs are observed in 2 or more of 6 subjects (or ≥33% of the cohort) at a dose level, the dose at which this occurs will be considered intolerable and the MTD will have been exceeded. The MTD is the dose below the intolerable dose.
  RP2D is the recommended Phase 2 dose, which was determined to be 80 mg
Time Frame: From time of first dose of PLX2853 and carboplatin until 30 days of end of treatment an average of 6 months.
Population: Note that the MTD was not reached as the study terminated early.
Measure: Count of Participants; unit: Participants
Groups:
- PLX2853 Phase 2a Monotherapy: Subjects with ARID1A mutation-positive advanced gynecological malignancies
Arm/Group | PLX2853 Phase 2a Monotherapy | PLX2853 + Carboplatin Phase 1b/2a Combination Therapy
Number analyzed (Participants) | 14 | 23
Participants | 0 | 0

3. Primary Outcome: Phase 2a (PLX2853 + Carboplatin Combination): Number of Participants Reaching ORR as Measured by RECIST v1.1
Description: Overall response rate as measured by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Time Frame: From 8 weeks of treatment with PLX2853 and Carboplatin (Cycle 3 Day 1; 28 days per cycle) until completion of long term follow-up, an average of 6 months.
Population: as for outcome 1
Arm/Group | PLX2853 Phase 2a Monotherapy | PLX2853 + Carboplatin Phase 1b/2a Combination Therapy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Through 30 days after last dose of study drug, an average of 6 months
Groups:
- PLX2853 + Carboplatin Phase 1b/2a Combination Therapy: Phase 1b (PLX2853 + carboplatin combination): Up to 15 evaluable subjects with platinum-resistant EOC will be enrolled.
  Phase 2a (PLX2853 + carboplatin combination): Up to 26 evaluable subjects with platinum-resistant EOC will be enrolled.
  PLX2853: PLX2853 tablets
  Carboplatin: Carboplatin IV injection, 5 mg•min/mL
Arm/Group | PLX2853 Phase 2a Monotherapy | PLX2853 + Carboplatin Phase 1b/2a Combination Therapy
All-Cause Mortality (participants affected / at risk) | 5/14 | 11/23
Serious Adverse Events (participants affected / at risk) | 6/14 | 10/23
Other Adverse Events (participants affected / at risk) | 14/14 | 20/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLX2853 Phase 2a Monotherapy (N=14) | PLX2853 + Carboplatin Phase 1b/2a Combination Therapy (N=23)
sepsis (Infections and infestations) | 1 (1) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
anemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
hepatic hematoma (Hepatobiliary disorders) | 1 (1) | 0 (0)
fatigue (General disorders) | 1 (1) | 0 (0)
large intenstinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
gastric haemmorhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
lethargy (Nervous system disorders) | 0 (0) | 1 (1)
obstruction gastric (Gastrointestinal disorders) | 2 (2) | 1 (1)
pneumonia (Infections and infestations) | 0 (0) | 1 (1)
procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
pyrexia (General disorders) | 0 (0) | 1 (1)
syncope (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLX2853 Phase 2a Monotherapy (N=14) | PLX2853 + Carboplatin Phase 1b/2a Combination Therapy (N=23)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 8 (8)
Alanine aminotransferase increased (Investigations) | 2 (2) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 6 (6) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Bilirubin increased (Investigations) | 3 (3) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 7 (7)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 7 (7)
Dizziness (Nervous system disorders) | 0 (0) | 4 (4)
Dysgeusia (Nervous system disorders) | 2 (2) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Fatigue (General disorders) | 7 (7) | 13 (13)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastroesophageal reflex disease (Gastrointestinal disorders) | 3 (3) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 5 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4) | 4 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 6 (6)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 5 (5)
Influenza like illness (General disorders) | 0 (0) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Lymphocyte count decreased (Investigations) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 11 (11) | 18 (18)
Neutrophil count decreased (Investigations) | 0 (0) | 4 (4)
Edema (General disorders) | 1 (1) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Platelet count decreased (Investigations) | 4 (4) | 16 (16)
Proteinuria (Renal and urinary disorders) | 1 (1) | 3 (3)
Pyrexia (General disorders) | 3 (3) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 4 (4)
Vomiting (Gastrointestinal disorders) | 6 (6) | 10 (10)
Weight loss (Investigations) | 2 (2) | 4 (4)
Decreased white blood cell (Investigations) | 0 (0) | 5 (5)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Ascites (Gastrointestinal disorders) | 2 (2) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Vision blurred (Eye disorders) | 1 (1) | 2 (2)
Cystitis (Infections and infestations) | 2 (2) | 0 (0)
Eructation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Activated patrial thromboplastin time prolonged (Investigations) | 1 (1) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Upper airway cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dermatitis acneform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was discontinued early due to a business decision by the sponsor. Only combined data were provided for the combo arm. No outcome measures were evaluated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-03): https://cdn.clinicaltrials.gov/large-docs/19/NCT04493619/Prot_SAP_001.pdf